CLINICAL TRIAL: NCT03844737
Title: Evaluation of the VisuXL® Performance on Ocular Surface Discomfort, in Professional Water-polo Athletes Exposed to Pool Water for Prolonged Periods
Brief Title: Evaluation of the VisuXL® Performance on Ocular Surface Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VISUfarma SpA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VF-OS-003/2018
Record Dates: First submitted 2019-01-31; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Ocular Discomfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VisuXL® Treatment (Experimental)
  Interventions: Device: VisuXL®

INTERVENTIONS:
Device: VisuXL® — Treatment of discomfort forms of the ocular surface, in professional water-polo athletes exposed to pool water for prolonged periods.

SUMMARY:
VisuXL® is a medical device that is effective in various ocular surface disorders (ocular dryness, changes in the continuity of the corneal and conjunctival surface, environmental stress, exposure to UV and ionizing radiation, prolonged use of videoterminals, etc.). Therefore, the aim of this study is to demonstrate that the clinical benefits and quality of life of the swimmers, exposed for a long time to water added with chlorine, are strongly linked to the unique composition of the long-term VisuXL® medical device.

DETAILED DESCRIPTION:
This is a post-market, monocentric, open-label, randomized study of superiority, with the untreated eye considered as a comparator for the eye treated with VisuXL®, to demonstrate the effectiveness of VisuXL® in professional water-polo athletes exposed to pool water after VisuXL® ocular instillations for 2 months. Considered the category of subjects to study, the study is to be considered a fact-finding pilot study in a particular category of subjects.

The study population will be enrolled only after having signed the informed consent; in each enrolled subject, only one eye will be treated with VisuXL®, while the other no, as will be considered the comparator, so the two randomized groups will be divided by treated eyes:

* Untreated control eye
* Eye treated with VisuXL®

Each enrolled subject will be instructed to instill, TID, 1-2 drops of VisuXL® always in the same eye during the entire study, according to the present modality:

* Morning
* Before training (at least one hour before entering the pool)
* After training (maximum one hour after the end of the activity) Subjects will continue to instil 1-2 drops of VisuXL®, TID, always in the same eye, even in days without training (including weekends).

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged 14 to 33 years
2. Schirmer test I> 10 mm at 5 '
3. Willingness to participate in the study and possibility to sign the ICF; for athletes aged <18 years: parents' agreement for the participation of the child in the study
4. Discomfort of the ocular surface

Exclusion Criteria:

1. Pathologies of the anterior segment
2. Diagnosis of autoimmune diseases (eg SEL, Sjogren)
3. Diagnosis of metabolic diseases (eg diabetes, thyroid malfunction/disorder)
4. Entropion
5. Trichiasis
6. Deficiency of androgens sex hormones
7. Taking medications that can interfere with the secretion of the lacrimal gland
8. Connective tissue disease
9. Prior eye surgery
10. Hypersensitivity to the active ingredients contained in VisuXL®
11. Use of artificial tears in the 15 days before the start of the study

Ages: 14 Years to 33 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
break-up time (BUT) | measured at week 1, 2, 4 and 8 versus baseline
  change over time in tear film break-up time (BUT)

SECONDARY OUTCOMES:
coloration of the ocular surface | measured at week 1, 2, 4 and 8 versus baseline
  Analysis to evaluate the differences over time between the two groups on coloration of the ocular surface (corneal and conjunctival) with fluorescein
Schirmer I test at 5 min (ST) (without anesthesia) | measured at week 1, 2, 4 and 8 versus baseline
  Analysis to evaluate the differences over time between the two groups on Schirmer I test at 5 min (ST) (without anesthesia)
Number of beating of eyelashes per minute | measured at week 1, 2, 4 and 8 versus baseline
  Analysis to evaluate the differences over time between the two groups on number of beating of eyelashes per minute
Tear osmolarity test | measured at week 1, 2, 4 and 8 versus baseline
  Analysis to evaluate the differences over time between the two groups on tear osmolarity test
Evaluation of visual acuity | measured at week 1, 2, 4 and 8 versus baseline
  Analysis to evaluate the differences over time between the two groups on evaluation of visual acuity
Questionnaire scores (OSDI) | measured at week 1, 2, 4 and 8 versus baseline
  Analysis to evaluate the differences over time between the two groups on questionnaire scores (OSDI). The overall Ocular Surface Disease score defined the ocular surface as normal (0-12 points) or as having mild (13-22 points), moderate (23-32 points), or severe (33-100 points) disease.
Subject satisfaction (10 points on the VAS scale) | measured at week 1, 2, 4 and 8
  Analysis to evaluate the differences over time between the two groups on subject satisfaction.
  (VAS: scale where patient has to specify level of satisfaction by indicating a position along a continuous line between two end-points (0 - 10). 0 indicates no satisfaction while 10 represents the highest level).

CONTACTS AND LOCATIONS:
Locations (1):
- UO Oculistica, Fondazione Policlinico Universitario A. Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided